CLINICAL TRIAL: NCT02196454
Title: Educating Pre/Teens and Their Parents on the Importance of HPV Vaccination
Brief Title: Video to Promote HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Noble Medical, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 14-011091
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Vaccine Acceptance; Social Acceptance; Acceptance Processes; Health Behavior; Human Papillomavirus
Keywords: HPV vaccine; vaccination; immunization; video; health education; communication
MeSH Terms: conditions — Behavior; Health Behavior; Health Education; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine Information Statement (No Intervention): Study participants will receive the HPV Vaccine Information Statement (VIS) which is part of routine care.
- Video & Vaccine Information Statement (Experimental): Participants will view an educational video about the HPV vaccine with a male or female narrator. Participants will also receive the HPV Vaccine Information Statement (VIS) which is part of routine care.
  Interventions: Other: Educational Video with Male or Female Narrator

INTERVENTIONS:
Other: Educational Video with Male or Female Narrator — Participants will watch an educational video about the quadrivalent HPV vaccine (Gardasil) narrated by either a male or female.
  Arms: Video & Vaccine Information Statement

SUMMARY:
The purpose of this research study is to determine if video-based education will increase HPV vaccination rates among 11 - 17 year olds.

DETAILED DESCRIPTION:
Human Papillomavirus (HPV) is a common sexually transmitted infection that has the potential to cause cancer. The vaccine is recommended because it prevents the HPV infections that most commonly cause cancer. HPV vaccines offer the best protection to girls and boys who receive the complete, three-vaccine series and have time to develop an immune response before being exposed to HPV. However, vaccination rates are low compared to other vaccines for teens.

Results from this study will help us learn why participants do or do not get the HPV vaccination and whether video-based education can help improve vaccination rates

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyads in which the child is a male or female age 11 to 17 years who has not received the HPV vaccine

Exclusion Criteria:

* Parent-child dyads in which the child has received the HPV vaccine
* Parent-child dyads in which the child is older than 18 at the time of enrollment
* Non-English speakers

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
HPV Vaccination Series Initiation | 90 days
  Number of HPV vaccine doses received among study participants
HPV Vaccine Series Initiation | 0 days
  HPV Vaccine Receipt among study participants

SECONDARY OUTCOMES:
HPV Vaccine Series Initiation (depending on male versus female narrator) | 0 days
  Difference in rate of HPV vaccine receipt between study participants who viewed a video narrated by a male versus a female
HPV Vaccine Series Initiation (depending on male versus female narrator) | 90 days
  Difference in number of HPV vaccine doses between study participants who viewed a video narrated by a male versus a female

OTHER OUTCOMES:
HPV Vaccine Awareness | 0 days
  Reported reason for HPV vaccine receipt or deferral

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A. Feemster, MD MPH MSHP, Principal Investigator — Children's Hospital of Philadephia
Locations (2):
- United States (2):
  - Primary Care, Flourtown, Children's Hospital of Philadelphia, Flourtown, Pennsylvania
  - Nicholas and Athena Karabots Pediatric Care Center, Philadelphia, Pennsylvania